CLINICAL TRIAL: NCT02103920
Title: A Retrospective Immunohistochemistry Study of the Expression of Glycine/ Serine Pathway Molecules in Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: MC01/06/11
Record Dates: First submitted 2012-04-02; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Solid Tumor Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the expression of molecules involved in the glycine/serine pathway using immunohistochemistry in solid tumors. Archived paraffin-embedded pathological specimens from the Department of Pathology, NUH will be obtained. Tissue microarray (TMA) is a high-throughput method of analysing large numbers of formalin-fixed, paraffin-embedded tumor at a minimal cost and effort. To analyse the expression of molecules of putative relevance to the glycine/serine pathway, (such as PSPH, PSAT1, SHMT1, and GLDC), TMA technology will be utilised as previously reported (Kristiansen, Zhang, Soong). Tissue arrays will be constructed from solid tumors including cancers of the colon/ rectum, lung, breast, cervix, ovary, endometrium, fallopian tube, prostate, kidney, testis, stomach, liver, brain and lymphoma. One hundred cases of each tumor type (subject to availability) will be stained using immunohistochemistry. Patient Identifiers will not be collected. Societal benefit in terms of knowledge gained to improve understanding of cancer. No direct risk to subjects as this is a retrospective study of archived pathological tumour samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumor cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Archived paraffin-embedded pathological specimens from the Department of Pathology, NUH.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change the expression of molecules of putative relevance to the glycine/serine pathway | 5 years
  Archived paraffin-embedded pathological specimens from the Department of Pathology, NUH will be obtained. Tissue microarray (TMA) is a high-throughput method of analysing large numbers of formalin-fixed, paraffin-embedded tumor at a minimal cost and effort. To analyse the expression of molecules of putative relevance to the glycine/serine pathway, (such as PSPH, PSAT1, SHMT1, and GLDC), TMA technology will be utilised as previously reported (Kristiansen, Zhang, Soong). Tissue arrays will be constructed from solid tumors including cancers of the colon/ rectum, lung, breast, cervix, ovary, endometrium, fallopian tube, prostate, kidney, testis, stomach, liver, brain and lymphoma. One hundred cases of each tumor type (subject to availability) will be stained using immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore